CLINICAL TRIAL: NCT06125626
Title: Prevention of Traveler's Diarrhea While Crossing the Amazon Forest by Bike With a Supplement Based on Lacticaseibacillus Rhamnosus LR04 + Streptococcus Thermophilus FP4 + Bifidobacterium Brevis BR03: a Phase Two, Randomized, Placebo-controlled, Double-blind, Cross-over Pilot Study
Brief Title: Prevention of Traveler's Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Nicola Veronese, Professor, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 153/2023
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): This arm will receive a daily sachet of Lacticaseibacillus rhamnosus LR04 + Streptococcus thermophilus FP4 + Bifidobacterium breve BR03
  Interventions: Dietary Supplement: Probiotical
- Placebo (Placebo Comparator): This arm will receive a dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotical — A daily sachet of Lacticaseibacillus rhamnosus LR04 + Streptococcus thermophilus FP4 + Bifidobacterium breve BR03 will be given to this group
  Arms: Probiotics
Other: Placebo — A daily sachet of placebo will be given to this groups
  Arms: Placebo

SUMMARY:
The prevention of traveller's diarrhea makes use of the selection of foods and drinks, the purification of water, the use of pharmacological substances such as bismuth salicylate and rifaximin (which can only be taken for short periods). The very attractive prospect of preventing travellers' diarrhea without systemic antibiotics has fueled interest in probiotics for this purpose. However, not all probiotics are identical, and the results of studies conducted with a particular agent cannot be generalized to indicate that any probiotic agent would be successful in the same clinical situation. Probiotics such as Lactobacillus GG have been shown to reduce the incidence of diarrhea in travelers in randomized controlled trials. In contrast, another Lactobacillus preparation, non-viable Lactobacillus acidophilus, showed no benefit over placebo in a randomized, double-blind, controlled trial of 174 travelers. The reasons for this are unclear, but could be related to the fact that the bacteria were not viable or a peculiarity of the strain selected for testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy bikers
* Able to pass the Amazonia forest by bike

Exclusion Criteria:

* None predifinied

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | 12 weeks
  Diarrhea will be defined using the Bristol's scale (value of 7) in a scale between 1 and 7, higher values reflecting more diarrhoic attitude

SECONDARY OUTCOMES:
Mean quality of life | 12 weeks
  Quality of life will be assessed using the short-form 12 (SF-12) with a standardized score between 0 and 100% compared to the Italian population.
Incidence of severe diarrhea | 12 weeks
  Severe diarrhea will be defined as a diarrhea requiring hospitalization or intravenous hydratation

CONTACTS AND LOCATIONS:
Locations (1):
- Nicola Veronese, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.iosonoamazzonia.org/it/temporary-home/

REFERENCES:
- [Background] Briand V, Buffet P, Genty S, Lacombe K, Godineau N, Salomon J, Vandemelbrouck E, Ralaimazava P, Goujon C, Matheron S, Fontanet A, Bouchaud O. Absence of efficacy of nonviable Lactobacillus acidophilus for the prevention of traveler's diarrhea: a randomized, double-blind, controlled study. Clin Infect Dis. 2006 Nov 1;43(9):1170-5. doi: 10.1086/508178. Epub 2006 Sep 27. PMID 17029137
- [Background] Hilton E, Kolakowski P, Singer C, Smith M. Efficacy of Lactobacillus GG as a Diarrheal Preventive in Travelers. J Travel Med. 1997 Mar 1;4(1):41-43. doi: 10.1111/j.1708-8305.1997.tb00772.x. PMID 9815476